CLINICAL TRIAL: NCT06293222
Title: Patient and Public Involvement and Engagement in Research on Life-limiting Conditions With Children and Young People With Sickle Cell Disorder and Their Families
Brief Title: Patient and Public Involvement and Engagement in Research With Children and Young People With Sickle Cell Disorder and Their Families
Status: Active, not recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Sickle Cell Society (Unknown)
Responsible Party: Sponsor
Other Study IDs: SCD Support
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Participants with personal experience of sickle cell disorder.: Participants with personal experience of sickle cell disorder (parents, affected children or siblings).
- Researchers: Researchers working with children with life limiting or life changing conditions
- Members of a patient advocacy organisation: Members of a patient advocacy organisation (Sickle Cell Society)

SUMMARY:
Aim: To co-produce resources for inclusive and equitable Patient and Public Involvement and Engagement in research on life-limiting conditions, with children and young people with sickle cell disorder and their families.

Methods: Workshops with a) members of a patient advocacy organisation (Sickle Cell Society n=5) b): i) Children and young people (10-18 years) with sickle cell disorder (n=15) and ii) their siblings (10-18 years, n=10) and iii) their parents (n=15), c) Researchers form the Cicely Saunders Institute Outputs: Resources that enable children and young people with sickle cell disorder and their families to engage in research

DETAILED DESCRIPTION:
Aim:

To co-produce resources for inclusive and equitable Patient and Public Involvement and Engagement in research on life-limiting conditions, with children and young people with sickle cell disorder and their families.

Objectives:

1. Partner and collaborate with the Sickle Cell Society to continue to build on the work of the Cicely Saunders Institute to support a thriving Patient and Public Involvement and Engagement community that includes children and young people and their families
2. Listen, hear, and understand what is important for children and young people with sickle cell disorder and provide them with the knowledge and skills to collaborate with researchers at the Cicely Saunders Institute during the design and implementation, analysis, and publication of research
3. Equip staff within the Cicely Saunders Institute with the knowledge, understanding and awareness of the role children and young people with sickle cell disorder and their families can play in patient-involved research to ensure pathways for prioritizing and disseminating patient led research are realised
4. Use data from objectives 1-3 to co-produce resources that may be used with a broader population of children and young people with serious and life-limiting conditions and their families to enable them to become equal partners in research
5. Use learning from the proposed project with the Sickle Cell Society as an exemplar partnership, to inform future Patient and Public Involvement and Engagement with children and young people with other serious and life-limiting conditions including cancer and neuro-disabilities as the investigators expand the research remit at the Cicely Saunders Institute.

Background:

Public involvement must be diverse and inclusive to enable research that has the potential to reach those that stand to benefit from it the most, and thus to address issues of health equity and accessibility. Yet, long-standing evidence has shown that those most likely to be involved in research come from a narrow section of the population, from older age groups, white ethnic and higher socio-economic backgrounds. It is widely recognised that many groups are underserved and underrepresented in research.

Underserved groups include children, young people and adults from different minority ethnic groups, socio-economically disadvantaged groups, migrants, asylum seekers, people with mental health conditions and multiple health conditions. Children and young people, as a group have few opportunities for research involvement. There is also limited evidence on optimal models for partnerships in research.

Changing the balance of power and promoting wider participation, empowerment, diversity, and equality, are seen as neglected aspects of involvement that, if given due attention, can offer a way to move beyond involvement at the lowest levels of consultation to partnering and collaborating with a wider diversity of people and communities.

Methods:

Design: A sequential design involving three work packages

• WP1 will address Objectives 1 and 2: Apr-June 2023

The investigators will hold separate child and adult online/face to face scoping workshops (n=3) with:

Group B(i) children and young people with sickle cell disorder (n=15) and B(ii) their siblings (n=10) and B(iii) their parents (n=15) recruited via charity partners to:

(i) Explain what research is, how it is conducted, relevant policies and the mission statement of the Cicely Saunders Institute (ii) Review structures and processes for equitable and inclusive Patient and Public Involvement and Engagement for children and young people with sickle cell disorder and their families (iii) Identify relevant and appropriate training/education/skills needed to enable children and young people with sickle cell disorder and their families to engage in research.

The child and young people's workshop will be facilitated by an artist to assist with activities to engage participants. These workshops will be evaluated by those involved using surveys which will be administered at the end of the workshops.

* WP2 will address objective 3: Jul-Aug 2023 The investigators will hold online/face to face workshops (n=2) with researchers from the Cicely Saunders Institute (n=10) and members of Group B (n=10-15) to enable them to work together to identify resources needed for meaningful Patient and Public Involvement and Engagement with children and young people with sickle cell disorder and their families to take forward into WP3. These workshops will also be evaluated by those involved using surveys which will be administered at the end of the workshops.
* WP3 will address objectives 4 and 5: Sept-Dec 2023 Through a combination of online/face to face working groups (n=2), the investigators will work with children and young people with sickle cell disorder and their families (n=10-15 at each workshop) as well as researchers from the Cicely Saunders Institute (n=5) to co-produce resources that enable them to engage meaningfully in research incorporating the skills and knowledge identified in WP1. One of these workshops will be facilitated by an artist to help children develop their ideas into future resources for meaningful Patient and Public Involvement and Engagement. This will facilitate their involvement in future funding applications that are driven by them.

The investigators will have a final celebratory event with Group A: Sickle Cell Society and Groups B(i) children and young people with sickle cell disorder (n=15), Bii) their siblings (n=10) and Biii) their parents (n=15) to showcase achievements and plan next steps. The celebratory event will include an evaluation of the whole project.

Outputs:

WP1: (i) Partnership with a charity organisation, the Sickle Cell Society (ii) guidance on reaching minority ethnic groups and publicizing research opportunities; (iii) training skills analysis to enable children and young people with sickle cell disorder and their families to engage in research in a meaningful way.

WP2: Identification of resources needed to facilitate meaningful involvement of children and young people with sickle cell disorder and their families to engage in research WP3: (i) Resources that enable children and young people with sickle cell disorder and their families to engage in research (ii) a future strategy for meaningful Public Involvement and Engagement with children and young people with sickle cell disorder and their families (iii) an exemplar to inform future Patient and Public Involvement and Engagement with children and young people with other serious and life-limiting conditions including cancer and neuro-disabilities as the investigators expand the research remit.

ELIGIBILITY:
Inclusion Criteria:

* Group A: Members of a patient advocacy organisation (Sickle Cell Society n=5)
* Group B:

  i) Children and young people (10-18 years) with sickle cell disorder (n=15) ii) their siblings (10-18 years, n=10) iii) their parents (n=15)
* Group C: Researchers working with children with life-limiting or life changing conditions

Exclusion Criteria:

* Group A: Members of patient advocacy organisations other than the Sickle Cell Society
* Group B:

  i) Children and young people younger than ten years or older than 18 years and those without sickle cell disorder (n=15) ii) siblings younger than ten years or older than 18 years and without a brother or sister with sickle cell disorder iii) parents of children with conditions other than sickle cell disorder
* Group C: Researchers who do not have experience working with children with life-limiting or life changing conditions

Min Age: 10 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: * Group A: Members of a patient advocacy organisation (Sickle Cell Society n=5)
  * Group B:
    i) Children and young people (10-18 years) with sickle cell disorder (n=15) ii) their siblings (10-18 years, n=10) iii) their parents (n=15)
  * Group C: Researchers working with children with life-limiting or life changing conditions
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Workshops with participants to develop resources that enable children and young people with sickle cell disorder and their families to engage in research | 8 months
  Resources that enable children and young people with sickle cell disorder and their families to engage in research

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data from the study are likely to be made available on request from the CI. Data may not be publicly available due to ethical constraints.

REFERENCES:
- [Derived] Chudleigh J, Follett A, Mcfarlane-Griffith E, Abuo D, Josh, Imani, Holder P. Exploring How Children and Young People With Sickle Cell Disease and Their Families Want to be Involved in Research: A Qualitative Study. Health Expect. 2025 Apr;28(2):e70242. doi: 10.1111/hex.70242. PMID 40152512